CLINICAL TRIAL: NCT04516512
Title: SARS-CoV-2 Seroprevalence Among Adults People Living in Jail
Brief Title: Assessment of SARS-CoV-2 Seroprevalence in Detention
Acronym: COVIDET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: APHP200667
Record Dates: First submitted 2020-08-17; First posted 2020-08-18 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; inmates; seroprevalence
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigated arm (Experimental): Participants included in the study who met inclusion criteria
  Interventions: Biological: Blood draw

INTERVENTIONS:
Biological: Blood draw — For each participants to the research a peripherical blood draw will be performed

SUMMARY:
"Background France counted on January 1, 2020, 70,651 people detained, for 61,080 places. Overcrowding in detention is considered as risk factor for infectious diseases transmission, such as respiratory infections. The prison environment represents a confined environment, which could protect prisoners from possible external contamination. If one or more inmates were infected through visiting rooms, officers working in detention, or newly incarcerated people, an epidemic could spread more quickly in the prison community. Thus, few cases of COVID-19 were observed among the subjects in detention with a few weeks delay compared to the free world. However, detention conditions make it more difficult to detect suspicious cases. On the other hand, carrying out diagnostic tests is structurally more difficult to carry out there. Thus, given the plurality of clinical presentations, the non-optimal sensitivity of the SARS-CoV-2 RT-PCR, and the difficulty in carrying out diagnostic tests, it is today difficult to have a precise idea of the number of prisoners having encountered SARS-CoV-2. It is also a population that is not taken into account in the large seroprevalence studies currently conducted in the general population. In order to estimate the number of prisoners exposed to SARS-CoV-2 and in the absence of data currently available in the medical literature, a seroprevalence study in this at risk and little studied population would bring new data to the medical community.

Hypothesis In adult subjects living in penal establishments in Ile de France, the seroprevalence of SARS-CoV-2 would be lower compared to the general population.

Material and method Open multicenter cross-sectional study carried out in the 11 penal establishments of Ile de France. A sampling of 3,500 inmates stratified over the 16 detention areas concerned will be carried out. The inclusion criteria will be detained subjects who have expressed their consent to participate in the research, aged 18 to 80 years. Each selected detainee will be invited to the health unit to perform a venous blood test for anti-SARS-CoV-2 antibodies. The goal is to take 2,500 blood samples (30% expected refusal rate). Each sample will be analyzed in the virology laboratory at P. Brousse hospital.

Expected results Obtain an assessment of the seroprevalence of SARS-CoV-2 in prisons to determine the exposure of detained persons. This assessment will make it possible to undertake public health actions and to propose the implementation of group protection measures such as vaccination if this is soon available.

DETAILED DESCRIPTION:
"

1. Scientific justification for the research

   o Current knowledge

   SARS-CoV-2, a new coronavirus infecting human, is responsible for the COVID-19 pandemic. The virus is transmitted either directly through the projection of contaminated droplets during a cough or sneeze, or indirectly through contact via an inert contaminated surface. The recent occurrence of the COVID-19 epidemic and the originality of the situation, both nationally and internationally, do not currently allow data describing the epidemic in prison, nor elements characterizing it the seroprevalence of SARS-CoV-2 in detention.

   The medical literature currently reports some reflections on the challenges of SARS-CoV-2 infection in prisoners. A team recently reported an epidemic of COVID-19 in prison in China3, which involved more than 500 cases including male and female prison staff and detainees.

   A recent publication reported that the infectious period of SARS-CoV-2 begins two to three days before the onset of symptoms4. This major fact could limit the effectiveness of the strategy currently adopted in detention to isolate everyone as soon as the first symptoms of COVID-19 appear, even if all the identified contact subjects were also placed in containment and monitored and the new arrivals in detention placed in solitary confinement for a period of 14 days.

   On January 1, 2020, France had 70,651 people detained, for 61,080 places. This overcrowding is concentrated in certain prisons which house 2/3 of the prison population, so the occupancy rate can reach 138%, forcing two to three people - sometimes more - to share the same cell. Overcrowding and overcrowding in detention are considered to be risk factors for the transmission of infectious diseases compared to the open environment, in particular for respiratory viruses. Thus, epidemics of influenza have been reported there in the United States and recently epidemics of SARS-CoV-2 in China.

   Since January 24, 2020, the date on which a Chinese tourist visiting France was identified as the first case infected with SARS-CoV-2 on the territory, the epidemic has spread widely in the general population, putting in straining the healthcare system and having led to major decisions aimed at reducing its transmission. While on February 25 died the first French patient following a COVID-19, almost three weeks later died of this disease, the first patient detained. He had been incarcerated eight days earlier. The rapid spread of the epidemic in the free world and the occurrence of this first death in detention then raised fears of an epidemic in prison. However, the prison environment alone represents a confined environment, which could protect prisoners from possible external contamination. According to some authors, the attack rate varies according to the number of people living in ""closed societies"" and the nature of their interactions and is not different from that observed in the general population.

   To reduce the risk of detainees being exposed to SARS-CoV-2, measures such as the early release agreement, the reduction in the number of arrivals, and the suspension of visiting rooms have been put in place. Thus, the number of prisoners in French prisons decreased by 6,266 people between March 16 and April 1.

   Although these actions were put in place, measures to limit human-to-human contamination of SARS-CoV-2 were difficult to apply at the start of the epidemic in the absence of sufficient supplies. Thus, in certain detentions, several grouped cases of COVID-19 have been observed among caregivers and prison staff. It is not excluded that these agents could have contaminated detained persons who run the risk of being disseminated to the incarcerated population because of the existing promiscuity.

   A few confirmed cases of COVID-19 have thus been observed among subjects detained a few weeks late compared to the free world in penal establishments in Ile de France, which corroborates the fact that the virus is present and circulating in the prison community. However, conditions of detention make it more difficult to detect suspicious cases, since detainees do not wish to be stigmatized among their fellow prisoners, tend to minimize or conceal their symptoms and thus make it less easy to consult the detention health unit (medical service). On the other hand, carrying out diagnostic tests is structurally more complex. In addition, the plurality of clinical presentations, the sensitivity of the SARS-CoV-2 RT-PCR which does not exceed 70% 10, and the difficulty in carrying out diagnostic tests, does not allow a precise idea of the number of inmates who encountered SARS-CoV-2.

   o Research hypotheses

   The seroprevalence of SARS-CoV-2 would be lower in detention compared to the general population.

   o Description of the population to be studied

   Population of adult subjects detained in penal institutions in Ile-de-France. The characterization of this specific population is necessary in France because no study to date reports data concerning this fragile and confined population due to the conditions of detention. Ile-de-France is one of the two regions with the Great East most affected by SARS-CoV-2.
2. Research objectives

   o Main objective of the research

   The main objective of the research is to assess the prevalence of SARS-CoV-2 infection among subjects detained in penal institutions in Ile-de-France.

   o Secondary research objectives

   The secondary objectives are:
   * Compare this prevalence to that of the general population
   * Describe the clinical forms in prisoners with a positive SARS-CoV-2 serology
   * Describe the characteristics and co-morbidities associated with a positive SARS-CoV-2 serology in detained subjects.
   * Evaluate the perception of the risk, the knowledge of the barrier measures and the recourse to care in case of symptoms in the detained subjects.
3. Description of the research methodology

   o Experimental design

   This is a multi-center cross-sectional seroprevalence study.
   * Number of participating centers Eleven penal establishments in Ile de France. The subjects will be recruited from the health units of penal establishments in Ile de France. These health units are all attached to hospitals.
   * Sample design

   Unit investigated: individual aged 18 to 80 detained in one of the 16 detention areas of the eleven prison centers in Ile-de-France.

   Sample size: the calculation of the number of subjects required results in 2500 subjects, a sampling of 3600 prisoners will therefore be carried out by probabilistic survey from the lists of prisoners provided by each center taking into account a probable rate of refusal of participation or release from detention between selection and inclusion of 30% (observed in a previous study).
4. Research process 4.1.1 Research calendar

   * Maximum time between selection and inclusion: 4 months
   * Duration of the inclusion period: 4 months 4.1.2 Selection visit

   No selection visit will be made, each participant drawn will receive a letter explaining the purpose and course of this research and inviting him to participate, the study information note will be attached to this letter. The letter will include a reply coupon which will be sent by the participant to the health unit if he wishes to participate in the research. Subjects who have thus responded positively will be invited to go to the health unit for the inclusion visit. If the subject does not appear at the health unit after a first invitation, a second invitation will be sent to him, if this second invitation is not honored, the subject will not be included in the study.

   4.1.3 Inclusion visit
   * The inclusion of subjects will take place in the health units of penitentiary establishments during a medical consultation. This visit will be provided by a doctor from the health unit and a nurse. During this visit, the investigative team:
   * Check the inclusion and non-inclusion criteria.
   * Explains the objective and the course of the research and obtains the signed consent. If the participant does not understand French, the investigator uses a translator.
   * Performs physical and clinical examination
   * Collects demographic and medical history data.
   * Carries out an interrogation in connection with the COVID-19 disease: Interrogates the subject to gather information concerning the possible symptoms in connection with COVID-19 felt since the end of February, the recourse to possible care, the factors supposed in connection with the infection with SARS-CoV-2 and the occurrence of moderate to severe forms of COVID-19, then asked him questions about his fear of being infected, his knowledge of the transmission of the virus and the barrier measures to put in place.
   * Performs peripheral venous sampling.

   The pseudo-anonymized samples will be sent to the virology laboratory at Paul Brousse Hospital for serological tests and the constitution of the biological collection.

   For each patient, the virology laboratory will edit and transmit, via secure messaging to the investigative center, the report of the serology result with the identifier of the participant in the research.
5. Stopping rules 5.1.1 Criteria and methods for premature termination of participation in the search for a subject

   Any subject can stop participating in research and exit the study at any time and for any reason. The investigator may temporarily or permanently interrupt a subject's participation in the research for any reason that would best serve the subject's interests. In the event of premature termination of the search for a subject, or withdrawal of consent, the data concerning him collected before the premature termination may be used.

   5.1.2 How to replace these people, if applicable

   Subjects who prematurely stopped participating in the research will not be replaced.

   5.1.3 Stopping some or all of the research

   The promoter AP-HP reserves the right to definitively suspend the inclusions, at any time, if it turns out that the inclusion objectives are not met.

   Since the subjects 'participation period is less than one day, no arrangements for taking charge of subjects' follow-up will be put in place, in the event of premature cessation of research.
6. Effectiveness assessment

   o Description of the efficacy evaluation parameters

   The immunological analyzes will be carried out under the direction of Professor Roque-Afonso. The teams involved in this task are those of the virology laboratory at Paul Brousse Hospital.

   o Determination of immunological parameters

   Blood samples will be sent to the virology laboratory / CRB Paris-Sud by a dedicated transporter, these samples will be centrifuged and aliquoted and stored at -80 ° C at CRB Paris-Sud. An aliquot will be used for the detection of anti-SARS-CoV-2 IgG by the SARS-CoV-2 IgG Reagent Kit test (Abbott Diagnostics) according to the manufacturer's recommendations.
7. Vigilance As part of this study, adverse events (serious or not) are not to be notified to the sponsor. Notification must be made as part of the vigilance implemented as part of the treatment."

ELIGIBILITY:
Inclusion Criteria:

* Detained woman appearing on the lists supplied by the penitentiary establishments or detained man drawn by lot from the lists supplied by the penitentiary establishments.
* Age from 18 to 80 years old.
* Free and informed consent signed."

Exclusion Criteria:

* Subject likely not to respect the terms of the study
* Persons who are placed under legal protection
* Person released from detention between the day of selection and the day of the planned consultation
* Person who are not attending the inclusion consultation after two invitations
* Patient who do not speaking French and are not accompanied by a translator
* Pregnant and lactating women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1044 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Determination of the immunological parameters (Immunoglobins G) of the SARS-CoV-2 infection | 7 days
  It's obtained from ELISA tests carried out on blood samples. A subject will be considered to have been infected with the SARS-CoV-2 virus if anti-SARS-CoV-2 IgGs are detected in his blood sample.

SECONDARY OUTCOMES:
Symptoms suggestive of COVID-19 | 7 days
  (fever or feeling of fever, headache, muscle aches and / or pain, cough, unusual breathing and / or shortness of breath, chest pain and / or tightness, rhinorrhea, nausea and / or vomiting, diarrhea, anosmia , ageusia, unusual tiredness), onset of hospitalization for COVID-19, onset of hospitalization in intensive care for COVID-19
Factors assumed to be related to infection with SARS-CoV-2 and the occurrence of moderate to severe forms of COVID-19 | 7 days
  age, smoking, cardiovascular history, diabetes, chronic respiratory disease, renal failure, active cancer, immunosuppression, hepatic cirrhosis , obesity, splenectomy, acute chest syndrome, sickle cell syndrome, taking chlorpromazine, number of inmates in the same cell, ward for vulnerable people, date of incarceration.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Mellon, MD,MPH, Study Director — Etablissement Public de Santé National de Fresnes, Service de Médecine; Anne Maie Roque-Afonso, MD, MPH, Study Chair — Hôpital Paul Brousse, Service de Virologie; Anne Dulioust, MD, PhD, Study Chair — Etablissement Public national de Fresnes, Service de Médecine
Locations (1):
- USMP, Le Kremlin-Bicêtre, France